CLINICAL TRIAL: NCT01007682
Title: Intrusive Reexperiencing: The Role of Working Memory Capacity and Thought Suppression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 192/09
Record Dates: First submitted 2009-10-28; First posted 2009-11-04 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Memory
Keywords: intrusive memories

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Screening for working memory capacity (No Intervention)
- Distressing movie (Experimental): A distressing movie is presented to two groups (one group with high and one group with low working memory capacity). For each of the two groups, half of the participants are instructed to suppress thoughts of the movies after viewing it, while the remaining participants are instructed to allow the occurrence of memories of the movie.
  Interventions: Other: Show distressing movie and tell half of the two study groups to suppress memories of the movie

INTERVENTIONS:
Other: Show distressing movie and tell half of the two study groups to suppress memories of the movie — A distressing movie is presented to two groups (one group with high and one group with low working memory capacity). For each of the two groups, half of the participants are instructed to suppress thoughts of the movies after viewing it, while the remaining participants are instructed to allow the occurrence of memories of the movie.
  Arms: Distressing movie

SUMMARY:
This study aims at identifying risk factors for the development of intrusive reexperiencing symptoms. In particular, the investigators examine the influence of working memory capacity and thought suppression on the occurrence of unpleasant memories of a negative experience.

Hypothesis: People with high working memory capacities (HWMC) are able to successfully suppress memories of an unpleasant experience (presentation of a distressing movie). In contrast, in people with low working memory capacities (LWMC), attempts to suppress memories of an unpleasant experience inadvertently lead to an increase of these memories.

Study phase one: Assessment of working memory capacity in 200 healthy participants by means of a computerized task. Selection of 50 participants with HWMC and of 50 participants with LWMC who participate in study phase two.

Study phase two: Presentation of a distressing movie and subsequent assessment of memories of the movie during several days in the daily life of participants. Comparison of 4 groups regarding the frequency of instructions in daily life:(group 1: HWMC participants who are instructed to suppress thoughts of the movie, group 2: LWMC participants who are instructed to suppress thoughts of the movie, group 3: HWMC participants who are instructed to allow the occurence of thoughts of the movie, group 4: LWMC participants who are instructed to allow the occurence of thoughts of the movie)

ELIGIBILITY:
Inclusion Criteria:

* Older than 17 years

Exclusion Criteria:

* Insufficient knowledge of the German language, for the distressing movie arm of the study: Elevated levels of depression or posttraumatic stress symptoms prior to viewing of the distressing movie

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Number of intrusive memories | during one week after viewing the distressing movie

CONTACTS AND LOCATIONS:
Overall Officials: Monique C Pfaltz, PhD, Principal Investigator — Harvard University, Department of Pysychology; Jürgen Margraf, Prof, Study Chair — University of Basel, Department for Clinical Psychology and Psychotherapy
Locations (1):
- Harvard University, Department of Psychology, Cambridge, Massachusetts, United States